CLINICAL TRIAL: NCT04480502
Title: ENVASARC: A Pivotal Trial Of Envafolimab, And Envafolimab In Combination With Ipilimumab, In Patients With Advanced Or Metastatic Undifferentiated Pleomorphic Sarcoma Or Myxofibrosarcoma Who Have Progressed On Prior Chemotherapy
Brief Title: ENVASARC: Envafolimab And Envafolimab With Ipilimumab In Patients With Undifferentiated Pleomorphic Sarcoma Or Myxofibrosarcoma
Acronym: ENVASARC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN035SAR201
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Undifferentiated Pleomorphic Sarcoma; Myxofibrosarcoma
Keywords: sarcoma
MeSH Terms: conditions — Histiocytoma, Malignant Fibrous; Dermatofibrosarcoma; Sarcoma | interventions — envafolimab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): Patients treated with 300 mg of single agent envafolimab every three weeks
  Interventions: Biological: Envafolimab
- Cohort B (Experimental): Patients treated with envafolimab in combination with ipilimumab. Envafolimab will be given at 300 mg every three weeks. Ipilimumab will be given at 1 mg/kg every three weeks for a total of four doses.
  Interventions: Biological: Envafolimab; Drug: Ipilimumab
- Cohort C (Experimental): Patients treated with 600 mg of single agent envafolimab every three weeks
  Interventions: Biological: Envafolimab
- Cohort D (Experimental): Patients treated with envafolimab in combination with ipilimumab. Envafolimab will be given at 600 mg every three weeks. Ipilimumab will be given at 1 mg/kg every three weeks for a total of four doses.
  Interventions: Biological: Envafolimab; Drug: Ipilimumab

INTERVENTIONS:
Biological: Envafolimab — PD-L1 single domain antibody for subcutaneous injection.
  Other Names: KN035
Drug: Ipilimumab — CTLA-4 monoclonal antibody
  Other Names: Yervoy
  Arms: Cohort B; Cohort D

SUMMARY:
This is a multicenter open-label, randomized, non-comparative, parallel cohort pivotal study of treatment with envafolimab (cohort A and C) or envafolimab combined with ipilimumab (cohort B and D) in patients with locally advanced, unresectable or metastatic undifferentiated pleomorphic sarcoma (UPS)/myxofibrosarcoma (MFS) who have progressed on one or two lines of chemotherapy.

DETAILED DESCRIPTION:
This is a multicenter open-label, randomized, non-comparative, parallel cohort pivotal study of treatment with envafolimab (cohort A and C) or envafolimab combined with ipilimumab (cohort B and D) in patients with locally advanced, unresectable or metastatic UPS/MFS who have progressed on one or two lines of chemotherapy. Patients were previously assigned at random into one of two cohorts: cohort A of 80 patients who received single agent envafolimab (300 mg every 3 weeks by subcutaneous (SC) injection) or cohort B of 80 patients who received envafolimab (300 mg every 3 weeks by SC injection) in combination with ipilimumab (1 mg/kg every 3 weeks intravenously for four doses). Following amendment #3, patients will be assigned at random into one of two cohorts: cohort C of 80 patients who will receive single agent envafolimab (600 mg every 3 weeks by subcutaneous (SC) injection) or cohort D of 80 patients who will receive envafolimab 600 mg every 3 weeks by SC injection) in combination with ipilimumab (1 mg/kg every 3 weeks intravenously for four doses). Following amendment #4, enrollment into cohort D was terminated and no further interim analyses will be conducted on this cohort.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic undifferentiated pleomorphic sarcoma (UPS) or grade ≥ 2 myxofibrosarcoma (MFS)
* Documented progression following systemic chemotherapy
* At least one measurable lesion
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Adequate hematologic and organ function

Exclusion Criteria:

* More than two prior lines of chemotherapy for UPS/MFS
* Prior immune checkpoint inhibitor or immunomodulatory therapy
* Active autoimmune disease that has required systemic treatment
* Major surgery within 4 weeks of dosing of investigational agent
* Active additional malignancy
* Pericardial effusion, pleural effusion, or ascites
* Central nervous system metastases and/or carcinomatous meningitis
* Active hepatitis or cirrhosis
* Interstitial lung disease
* Unwilling to apply highly effective contraception during the study
* Other concurrent severe and/or uncontrolled medical conditions that would, in the investigator's judgment, contraindicate patient participation in the clinical study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 assessed by blinded independent central review | 40 months

SECONDARY OUTCOMES:
Duration of response (DR) assessed by blinded independent central review | 40 months
Disease control rate (DCR) assessed by blinded independent central review | 40 months
Progression free survival (PFS) assessed by blinded independent central review | 40 months
Overall survival (OS) | 40 months
Characterize envafolimab pharmacokinetics (PK) in patients receiving envafolimab as a single agent and in combination with ipilimumab | 40 months
Characterize ipilimumab PK in patients given ipilimumab with envafolimab | 40 months
Objective response rate (ORR) by investigator assessment | 40 months
Progression free survival (PFS) by investigator assessment | 40 months
Characterize the immunogenicity of envafolimab and ipilimumab | 40 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles Theuer, MD, PhD, Study Director — Tracon Pharmaceuticals Inc.
Locations (30):
- United States (29):
  - University of Arizona, Tucson, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Evanston, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - University Hospitals, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University (Sidney Kimmel Cancer Center), Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College of Wisconsin, Wauwatosa, Wisconsin
- Royal Marsden, London, United Kingdom